CLINICAL TRIAL: NCT06896227
Title: Transcatheter Aortic Valve Implantation (TAVR): The Impact of Prothesis Positioning on Valvular and Coronary Hemodynamics
Brief Title: TAVR: The Impact of Prothesis Positioning on Valvular and Coronary Hemodynamics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CaS
Record Dates: First submitted 2025-03-13; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-10

CONDITIONS: Transcatheter Aortic Valve Replacement; Transcatheter Aortic Valve Implantation; Commissural Alignment; Commissural Misalignment; Symmetry; Prothesis Positioning; Prosthesis Durability; Aortic Valve Stenosis; Aortic Valve Disease
Keywords: TAVR; TAVI; Commissural alignment; Symmetry; Prothesis positioning; cMRI; 4D Flow; TEE
MeSH Terms: conditions — Prosthesis Failure; Aortic Valve Stenosis; Aortic Valve Disease | interventions — Echocardiography; Echocardiography, Transesophageal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TTE, TEE and MRI after TAVR (Other): Each study patient will undergo transthoracic echocardiography, transesophageal echocardiography, and cardiac magnetic resonance imaging following transcatheter aortic valve replacement.
  Interventions: Diagnostic Test: transthoracic echocardiography

INTERVENTIONS:
Diagnostic Test: transthoracic echocardiography — Each study patient will undergo transthoracic echocardiography, transesophageal echocardiography, and cardiac magnetic resonance imaging following transcatheter aortic valve replacement.
  Other Names: Transoesophageal echocardiography; cardiac magnetic resonance imaging

SUMMARY:
The aim of this clinical study is to learn more about the effects of TAVR-prosthesis positioning on hemodynamics and the coronary arteries.

The main questions it aims to answer are:

1. Does the cardiac magnetic resonance imaging and the echocardiography imaging provide an equivalent alternative to the computer tomography which is the state of the art in evaluating commissural alignment?
2. What effect does the position of the valve on the annular level have, especially its symmetrical and commissural position, on valvular and aortic blood flow characteristics?
3. What is the influence of symmetrical position and the presence of a commissural alignment on the coronary flow after transcatheter aortic valve replacement?

DETAILED DESCRIPTION:
Coming from a treatment option only for a high-risk cohort of elderly patients, transcatheter aortic valve replacement (TAVR) has become a safe and effective therapeutic approach for most patients with severe aortic valve stenosis (AS). Therefore, current guidelines recommend TAVR in patients from the age of 75 and even low surgical risk. Especially with the increasingly younger patient clientele, lifetime management is of utmost importance. Lifetime management includes, for example:

* Preserving coronary access after TAVR
* "Durability" of the new valve.
* Prevention of paravalvular leakage
* Prevention of atrioventricular blocks, which may necessitate a pacemaker.

The first two factors are particularly important and have therefore become the focus of the work.

Relating to this, the investigators would like to investigate three points:

1. Coronary access after TAVR is an important aspect for especially younger patients with longer life expectancy. The manufacturers try to address this task by offering techniques, which should help to orientate the novel commissures of the TAVR-valve within the native commissures of the diseased valve. Until now, the commissural alignment (CA) or misalignment (misCA) can only be depicted by post-TAVR cardiac computer tomography (CT) or selective coronary angiography, coming along with additional radiation and contrast medium exposure. Cardiovascular magnetic resonance imaging (CMRI) as well as transoesophageal echocardiography (TEE) may be alternative diagnostic options but have not been tested so far.
2. Transvalvular blood flow characteristics depending on the position of TAVR-prosthesis at the annular level may play a significant role concerning prothesis durability. However, it is unknown whether an asymmetric position or the presence of a CA may alter flow profile and therefore cause secondary endothelial stress leading to long term damage. With transthoracic echocardiography (TTE), TEE and CMRI the investigators would like to characterize flow patterns depending on symmetric vs. asymmetric valve position and CA vs. misCA.
3. It is not known what influence the TAVR position, more precisely a symmetric implantation and the presence of a CA, has on coronary flow and clinical outcomes. To investigate this, the investigators will record coronary flow in TEE and CMR after the implantation.

The results could be used in the future to detect CA or misCA and thereby evaluate and improve implantation techniques without harming the patient. Furthermore, if the investigators can identify advantages in symmetrically implanted TAVR with CA in terms of valve and coronary flow, techniques can be developed that target both symmetric and CA.

ELIGIBILITY:
Inclusion Criteria

- Patients who have undergone transfemoral transcatheter aortic valve replacement (TAVR).

Exclusion Criteria

* Any access route other than transfemoral.
* Valve-in-valve procedures.
* History of prior bioprosthetic valve implantation.
* Presence of pacemaker, implantable cardioverter-defibrillator (ICD), or cardiac resynchronization therapy (CRT) system.
* Diagnosis of liver cirrhosis.
* Esophageal disorders, including but not limited to esophageal varices.
* Thrombocytopenia or coagulation disorders.
* Any medical or psychiatric condition (e.g., dementia, alcoholism, or substance abuse) that may impair the ability to provide informed consent or interfere with study procedures, including follow-up visits.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Presence of a commissural alignment | Day 1
  by transoesophageal echocardiograpy and cardiac magnetic resonance imaging
Presence of symmetrical position | Day 1
  by transoesophageal echocardiograpy and cardiac magnetic resonance imaging
Transvalvular gradients | baseline + day 1
  by Transthoracic echocardiography
Effective orifice area (EOA) | baseline + day 1
  by Transthoracic echocardiography
Doppler velocity index | baseline + day 1
  by Transthoracic echocardiography
Paravalvular leakage | Day 1
  by transoesophageal echocardiograpy
Turbulent flow | baseline + day 1
  by transoesophageal echocardiograpy and cardiac magnetic resonance imaging
Pressure recovery | Day 1
  by cardiac magnetic resonance imaging
Energy loss coefficient | Day 1
  by transoesophageal echocardiograpy
global coronary flow reserve | Day 1
  by cardiac magnetic resonance imaging
Peak velocity | Day 1
  by cardiac magnetic resonance imaging
Wall sheer stress | Day 1
  by cardiac magnetic resonance imaging
Flow displacement | Day 1
  by cardiac magnetic resonance imaging
aortic area | Day 1
  by cardiac magnetic resonance imaging
volumen | Day 1
  by cardiac magnetic resonance imaging
LV-Function | baseline + day 1
  by transthoracic echocardiograpy and cardiac magnetic resonance imaging
RV-Function | baseline + day 1
  by transthoracic echocardiograpy and cardiac magnetic resonance imaging
Strain | Day 1
  by transthoracic echocardiograpy

CONTACTS AND LOCATIONS:
Overall Officials: Malte Kelm, Prof., Study Chair — Division of Cardiology, Pulmonary Disease and Vascular Medicine; Tobias Zeus, Prof., Study Director — Division of Cardiology, Pulmonary Disease and Vascular Medicine; Kathrin Klein, Dr. med., Study Director — Division of Cardiology, Pulmonary Disease and Vascular Medicine
Locations (1):
- Division of Cardiology, Pulmonary Disease and Vascular Medicine at University Hospital Duesseldorf, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: No